CLINICAL TRIAL: NCT05875441
Title: A Phase 2, Placebo-controlled, Double-blind, Randomized, Dose Ranging, Efficacy and Safety Study of Orally Administered Moxidectin in Adults With Scabies.
Brief Title: Efficacy and Safety Study of Moxidectin in Adults With Scabies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDGH-MOX-2002
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Scabies
Keywords: Moxidectin; Oral
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized, dose ranging study. Four cohorts of 50 subjects per cohort are planned. Subjects will be randomized 1:1:1:1 to receive Moxidectin 8mg, Moxidectin 16mg, Moxidectin 32mg or Placebo as a single oral dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded. Subjects will be randomized to one of the treatment arm by Interactive Response Technology at 1:1:1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Moxidectin 8mg (Experimental): Moxidectin 8 mg (over encapsulated) will be administered as a single dose on Day 0. Each subject will receive the same number of capsules made up of moxidectin 2 mg over encapsulated tablets and placebo capsules to maintain the blind.
  Interventions: Drug: Moxidectin Oral Product
- Moxidectin 16mg (Experimental): Moxidectin 16 mg (over encapsulated) will be administered as a single dose on Day 0. Each subject will receive the same number of capsules made up of moxidectin 2 mg over encapsulated tablets and placebo capsules to maintain the blind.
  Interventions: Drug: Moxidectin Oral Product
- Moxidectin 32mg (Experimental): Moxidectin 32 mg (over encapsulated) will be administered as a single dose on Day 0.
  Interventions: Drug: Moxidectin Oral Product
- Placebo (Placebo Comparator): 16 Placebo capsules will be administered as a single dose on Day 0.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxidectin Oral Product — The required number of moxidectin 2 mg tablet over encapsulated capsules will be administered as a single dose with placebo capsules to match as required
  Arms: Moxidectin 8mg
Drug: Moxidectin Oral Product — The required number of moxidectin 2 mg tablet over encapsulated capsules will be administered as a single dose with placebo capsules to match as required
  Arms: Moxidectin 16mg
Drug: Moxidectin Oral Product — The required number of moxidectin 2 mg tablet over encapsulated capsules will be administered as a single dose.
  Arms: Moxidectin 32mg
Drug: Placebo — 16 placebo capsules will be administered as a single dose.
  Arms: Placebo

SUMMARY:
Moxidectin is not approved to treat scabies in humans. The effective dose of moxidectin to treat scabies is not known. This study aims to assess the efficacy of a single administration of 8 mg, 16 mg, or 32 mg moxidectin per oral in achieving Scabies Complete Cure at Day 28. This study also aims to assess the safety of three strengths of single moxidectin doses in adults with scabies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Provided written informed consent.
3. Diagnosis of active scabies infestation confirmed by the presence of clinical signs and symptoms (evidence of burrows or typical inflammatory/noninflammatory lesions and pruritus) and either microscopic confirmation of scabies mite(s), ova or scybala by skin scraping or dermoscopy.
4. All female subjects of childbearing potential must agree to the use of a highly effective method of birth control until 16 weeks after administration of Investigational Product (IP).

Exclusion Criteria:

1. Diagnosis of crusted/Norwegian scabies or scabies presentation that, in the opinion of the Investigator, would require treatment with more than one standard of care treatment for scabies (e.g., scabies requiring concurrent topical and oral treatment).
2. History of chronic or recurrent dermatologic disease or skin conditions other than scabies that could interfere with the diagnosis of scabies and evaluation of cure.
3. Received any treatment with one or more scabicides within the 28 days prior to Screening, or between Screening and Baseline, including but not limited to permethrin, ivermectin, benzyl benzoate, sulfur, lindane, crotamiton, malathion, tea tree oil or spinosad.
4. Body mass index > 35 kg/m2.
5. Creatinine clearance < 30 mL/min (using Cockcroft-Gault equation).
6. Both total bilirubin >1.5 x upper limit of normal (ULN) and AST > ULN.
7. Abnormal and clinically relevant findings in hematology or biochemistry assessments at Screening, or in vital signs, 12-lead ECG, or physical examination at Screening and/or Baseline, that in the opinion of the Investigator would put the subjects at increased risk from participating in the study, confound study evaluations, or may interfere with study conduct.
8. Presence of any other clinically relevant condition, including infection, immunological disorder, malignant disease, and/or other underlying condition or circumstance at Screening or Baseline that in the opinion of the Investigator would put the subjects at increased risk from participating in the study, confound study evaluations, or interfere with the study conduct.
9. Use of topical steroids, systemic or high-dose inhaled corticosteroids (>500 µg per day of fluticasone propionate or equivalent for adults), or other immunomodulators within 14 days of Baseline.
10. Requiring ongoing treatment with, or received within 5 half-lives before Screening, any of the following medications that are clinical BCRP inhibitors: curcurmin (turmeric) supplements, cyclosporine A, darolutamide, eltrombopag, febuxostat, fostamatinib, rolapitant and teriflunomide.
11. Received an investigational agent within 28 days of Screening (or 5 half-lives of the investigational agent, whichever is longer).
12. Known or suspected hypersensitivity to macrocyclic lactones or excipients used in the formulation of moxidectin or ivermectin.
13. Known or suspected hypersensitivity to any of the components in permethrin 5% cream, to any synthetic pyrethroid or pyrethrin, or to the components of spinosad 0.9% topical suspension.
14. Known, suspected or at risk of Loa loa coinfection.
15. Difficulty swallowing tablets or capsules.
16. Pregnant or breastfeeding or planning to become pregnant from Screening until 16 weeks after treatment with IP.
17. Known or suspected alcohol or illicit substance abuse.
18. Unwilling, unlikely or unable to comply with all protocol specified assessments.
19. Previous enrolment in this study.
20. Previous moxidectin exposure within 6 months (5 half-lives) from Baseline.
21. Has household members who refuse or are unable to receive permethrin 5% cream treatment for scabies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Proportion of index subjects achieving complete cure (Efficacy) | 28 Days
  Proportion of index subjects achieving Complete Cure at Day 28. Complete Cure is defined as demonstration of both:
  1. Clinical cure: all signs and symptoms have completely resolved, including burrows, inflammatory/noninflammatory lesions and pruritus. And
  2. Microscopic or dermatoscopic cure demonstrating the absence of mites, eggs, and/or scybala, and negative dermoscopy for burrows.
Incidence and severity of Treatment Emergent Adverse Event (Safety) | 84 Days
  Incidence and severity of Treatment Emergent Adverse Event (TEAEs), Incidence of serious TEAEs and Incidence of TEAEs leading to study withdrawal and/or death.

OTHER OUTCOMES:
Proportion of index subjects achieving clinical cure without microscopic or dermatoscopic cure, assessed by skin examination to confirm all signs of scabies have completely resolved. | 28 Days
  The proportion of index subjects demonstrating clinical cure without microscopic or dermatoscopic cure at Day 28.
Proportion of index subjects achieving microscopic or dermatoscopic cure without clinical cure. Microscopic or dermatoscopic cure is assessed by demonstrating the absence of scabies mites, eggs, and/or scybala, and negative dermoscopy for burrows. | 28 Days
  The proportion of index subjects demonstrating microscopic or dermatoscopic cure without clinical cure at Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Fernandez, MD, Principal Investigator — Advance Care and Clinical Trials; Jorge Lopez, MD, Principal Investigator — Hospital y Clinica Bendana; Daisy Blanco, MD, Principal Investigator — Instituto Dermatologico Dominicano y Cirugia de Pie; Jorge Castillo Molina, MD, Principal Investigator — Affinity Clinical Research Services; Patricia A Zuniga Munoz, MD, Principal Investigator — Derclinic; Laura B Vargas Rivas, MD, Principal Investigator — Vargas Clinic; Gilberto Perez, MD, Principal Investigator — Evolution Clinical Trials; Armando Pineda-Velez, MD, Principal Investigator — Medical Research of Westchester, Inc; Bruce Torkan, MD, Principal Investigator — LA Universal Research Center, Inc
Locations (9):
- United States (5):
  - LA Universal Research Center, Inc, Los Angeles, California
  - Evolution Clinical Trials, Miami, Florida
  - Advanced Care and Clinical Trials, LLC, Miami, Florida
  - Medical Research of Westchester, Inc, Miami, Florida
  - Affinity Clinical Research LLC, Tampa, Florida
- Instituto Dermatologico Dominicano y Cirugia de Piel, Santo Domingo Oeste, Santo Domingo Province, Dominican Republic
- Vargas Clinic, San Salvador, San Salvador Department, El Salvador
- Honduras (2):
  - Derclinic, San Pedro Sula, Cortez
  - Hospital y Clinica Bendana, San Pedro Sula, Cortés Department

IPD SHARING:
Plan to Share IPD: Undecided